CLINICAL TRIAL: NCT07313059
Title: Prospective Clinical Evaluation of Incidence, Outcomes and Individuals Experiences Following Diagnosis of Clonal Haematopoiesis in a Dedicated Research Clinic
Brief Title: CHAPTER: Clonal Haematopoiesis Assessment: Prevention, Treatment and Research
Acronym: CHAPTER
Status: Not yet recruiting | Type: Observational
Sponsor: Clinical Hub for Interventional Research (CHOIR) (Other Government)
Collaborators: Medical Research Future Fund (Other); Australian National University (Other); University of Auckland, New Zealand (Other); The Canberra Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 24-CH-001
Record Dates: First submitted 2025-11-26; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Clonal Hematopoiesis; CCUS Clonal Cytopenia of Undetermined Significance; Hematologic Disease and Disorders
Keywords: Clonal Hematopoiesis; CH; CCUS
MeSH Terms: conditions — Hematologic Diseases; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Peripheral blood research samples will be collected. After research samples have been processed, analysed, and stored for study endpoint evaluation, as specified in this protocol, the remaining specimens, if any, at the University of Auckland, if necessary. However, there is no long term dedicated storage of participant research samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
People identified to have CH or thought to have possible CH due to unexplained low blood cell counts, including low red blood cells, white blood cells, or platelets will be asked to take part in the study.

Individuals who are confirmed to have CH and provide informed consent to participate in the study will have monitoring of their CH, assessment of the risk of heart diseases, blood cancers and personalised support. The researchers will also measure people's understanding of CH and how they feel after learning about CH.

Researchers will then record the relevant information from people with CH in a central database over time to track long-term health outcomes.

The information collected from the study will help create a blueprint for doctors to provide care for people with CH in the future, and guide further research into CH in Australia.

Participants will be asked to donate blood samples for the study for research purposes including CH monitoring and testing and also provide health information for the central database.

DETAILED DESCRIPTION:
Clonal Haematopoiesis (CH) refers to the clonal outgrowth of a population of hematopoietic stem cells in the absence of haematologic neoplasms. The clonal cells share an acquired 'driver' mutation., and the presence of dysplasia and/or cytopenia.

CH is common in older populations, with a frequency of 10-30% in people above 70 years of age.

Most individuals with CH are asymptomatic; however, the condition increases the risk of multiple life-limiting complications, including myeloid neoplasms (MN), cardiovascular disease (CVD), cerebrovascular disease (CeVD) by 11.1, 1.4, and 2-fold, respectively. While CH is not yet treatable, identifying the condition may assist individuals in making informed decisions, including an individualised management plan for early detection of CH-associated complications. CH screening is not currently performed in routine clinical practice.

The optimal approach to surveillance for myeloid neoplasms in individuals with CH remains undefined. Some individuals undergo active surveillance with regular blood count monitoring to detect early progression to MN. Early detection of MN may also broaden the therapeutic window for individuals. Additionally, this allows individuals to connect with suitable clinical trials.

CVD is the most common CH-associated complication; hence CV (cardiovascular) risk modification is important both from an individual and public health standpoint.

CH screening may also refine the evaluation of individuals with unexplained cytopenia, as they may have underlying CH that has not been identified.

Given the uncertainties surrounding the identification and management, dedicated research clinics have been developed in the United States to evaluate the impact of screening of CH. These clinics provide a supportive environment to discuss the condition and engage multidisciplinary management. In addition to haematologists, individuals are supported by other specialities and allied health professionals. However, dedicated CH clinics are not yet available in Australia.

There is an urgent need for more research into CH as there are crucial knowledge gaps. This includes the role of CH screening and interventions to modify the biology and risks of CH-associated complications. Given the widespread use of next-generation sequencing (NGS) panels in Australia, it is likely that CH will be increasingly identified in routine clinical practice, creating a pool of individuals who may benefit from counselling and follow-up in a dedicated service.

This cohort study will establish a screening clinic and a prospectively characterised registry of individuals with CH to serve as the basis for clinical and translational studies in CH.

With consent, individuals with possible CH will undergo screening by molecular testing in the first dedicated multidisciplinary CH clinic in Australia whereby the health outcomes of participants with CH can be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 55 years and above
2. Confirmed CH or possible CH, with possible CH defined by:

   a. Persistent, non-severe cytopenia, characterised by one or more of the following, present on at least 2 occasions, at least 4 months apart: i. Absolute neutrophil count (ANC) < 1.8 x 109/L ii. Haemoglobin (Hb) < 115 g/L in females, < 135 g/L in males iii. Platelet count < 150 x 109/L
3. Provision of written informed consent prior to any study-related assessments or procedures being carried out.

Exclusion Criteria:

1. Severe cytopenia as defined by one or more of the following:

   1. ANC < 0.5 x109/L
   2. Hb < 80 g/L
   3. Platelet count < 50 x 109/L
2. Multilineage cytopenias:

   a. Marked trilineage cytopenia with all the following present: i. ANC < 1.0 x 109/L AND ii. Hb < 110 g/L AND iii. Platelet count < 100 x 109/L

   b. Marked bilineage cytopenia, with two or more of the following present: i. ANC < 1.0 x 109/L ii. Hb < 110 g/L iii. Platelet count < 100 x 109/L

   Note: People with possible CH, with the above characteristics will be excluded from referral to the CH clinic and will instead have urgent investigation as an inpatient or in the haematology clinic. However, if no definite cause for cytopenia is identified, including CH, then individuals may be referred for CH screening at the CH clinic the discretion of the study PI

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 55 years and over with confirmed CH (Group 1), and possible CH (Group 2) who meet the defined eligibility criteria. Around 100 participants will be recruited to the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2033-11 (Estimated); Study Completion 2033-11 (Estimated)

PRIMARY OUTCOMES:
Establishment of CH participant registry and characterisation of CH outcomes | Through study completion, 5 years

SECONDARY OUTCOMES:
Number and proportion of participants with CH in a population at risk | Through study completion, 5 years
Incidence of CH-associated complications | First Visit (Week 0), Second Visit (Week 6) and Follow Up Visits (Weeks 52, 104, 156, 208 and 260)
  The incidence of CH-associated complications will be measured by:
  A) The number and proportion of participants with CH-associated complications (i.e., MN, CVD, CeVD, thrombosis) B) The number and proportion of participants with high CVD risk, as assessed using AusCVDRisk, and modification in individuals with CH C) The number of CV risk factors in participants with CH
Number and proportion of participants with CH with good perception and quality of life | At Screening, Second Visit (Week 6) and Follow Up Visits (Weeks 52, 104, 156, 208 and 260)
  Individual's perception and understanding of CH changes over time will be measured and assessed using the Brief Illness Perception Questionnaire (B-IPQ)
Number and proportion of participants with CH with good understanding of the condition | Screening, Second Visit (Week 6) and Follow Up Visits (Week 52, 104, 156, 208 and 260)
  How an individuals' perception and understanding of CH changes over time will be measured using a custom CH survey
Number and proportion of participants with CH experiencing psychological distress | Screening, Second Visit (Week 6), Follow Up Visits (Week 52, 104, 156, 208, and 260)
  The prevalence of psychological distress in individuals with CH will be measured using the Kessler Psychological Distress Scale (K6)
Change in VAF in individuals with CH at different timepoints | Screening, Follow Up Visits (Week 52, 104, 156, 208 and 260)
  The changes in the VAF (Variant Allele Fraction) in individuals with CH over time will be measured biennially (every 2 years) in all individuals.
  DNA extracted from the peripheral blood will be sequenced after NGS library preparation and target-enrichment with a custom capture panel (Agilent Sure Select). Next Generation Sequencing (NGS) will be performed and the number of variant reads at a given position will be used to calculate the VAF. VAF will be a direct measure of the fraction of cells carrying the variant in the sample used for DNA extraction.
  High Risk - CH participants will have additional VAF testing at Week 104 and Week 208 only if indicated i.e. worsening cytopenia, concerning blood film features or development of CH-associated complication.
Morphological changes by morphological feature analysis of CH changes | First Visit (Week 0), Follow Up Visits (Week 52, 104, 156, 208 and 260)
  CH associated morphology changes on peripheral blood film appearance will be measured and analyzed using a computational method that detects and characterizes white and red blood cell features to identify CH-associated morphology features using deep learning approaches.
  Images of stained and unstained peripheral blood films, and associated data reports, will be collected from each participant for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Canberra Health Services, Canberra, Australian Capital Territory, Australia